CLINICAL TRIAL: NCT01343160
Title: Multicenter Study of Removable GORE VIABIL® Biliary Endoprosthesis for Treatment of Benign Biliary Strictures
Brief Title: Removable GORE VIABIL® Biliary Endoprosthesis for Treatment of Benign Biliary Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBR CS 156
Record Dates: First submitted 2011-02-14; First posted 2011-04-27 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Biliary Strictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GORE VIABIL® Biliary Endoprosthesis (Other): Placement of GORE VIABIL® Biliary Endoprosthesis to establish duct patency
  Interventions: Device: GORE® VIABIL® Biliary Endoprosthesis

INTERVENTIONS:
Device: GORE® VIABIL® Biliary Endoprosthesis — Deployment of GORE® VIABIL® Biliary Endoprosthesis to the area of stricture

SUMMARY:
The purpose of this study is to generate clinical data to support the use of GORE® VIABIL® Biliary Endoprosthesis in the endoscopic and percutaneous treatment of benign biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with treatable benign biliary stricture which necessitates the need for implantation of a biliary endoprosthesis
* Subject is ≥18 years of age
* Subject is able to comply with study protocol and follow-up requirements
* Written informed consent is obtained using the Investigational Review Board (IRB)/Ethics Committee (EC) approved consent form

Exclusion Criteria:

* Subject anatomy ruling out covered self expanding metal stent use (e.g. above hilar region)
* Treatment of stricture would require placement of a covered biliary endoprosthesis within a previously placed bare metal stent
* The subject has malignant biliary disease
* Subject has known pregnancy
* Participated in protocol involving investigational drug or device within 90 days prior to entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Caca, MD, Principal Investigator — Klinikum Ludwigsburg
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GORE VIABIL® Biliary Endoprosthesis
Started | 36
Completed | 31
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- GORE VIABIL: GORE® VIABIL® Biliary Endoprosthesis
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 07
  Male | 29
Region of Enrollment [Number; unit: participants]
  Germany | 33
  Belgium | 3

OUTCOME MEASURES:

1. Primary Outcome: Safe Stent Removal
Description: The stent removal is considered safe when the Study Device is removed successfully and without SAEs.
Time Frame: Upon Removal
Population: Subjects with stent removal data available
Measure: Count of Participants; unit: Participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 33
Participants | 33

2. Other Pre Specified Outcome: Primary Device Patency
Description: Primary device patency is defined as the freedom from device occlusion requiring intervention (during the treatment period).
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 36
percentage of participants | 77.7 [55.9 to 89.6]

3. Other Pre Specified Outcome: Successful Delivery and Deployment
Description: This requires successful delivery and deployment of the device at the intended site.
Time Frame: Upon Implant
Measure: Count of Participants; unit: Participants
Arm/Group | GORE VIABIL® Biliary Endoprosthesis
Number analyzed (Participants) | 36
Participants | 36

4. Other Pre Specified Outcome: Successful Treatment of Benign Stricture Upon Implant
Description: Successful treatment of strictures is defined as stricture resolution upon implant as reported by the PI. For the purpose of this report, we will be referring to this as "stented stricture resolution".
Time Frame: Upon implant
Measure: Number; unit: participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 36
participants | 35

5. Other Pre Specified Outcome: Secondary Patency
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 36
percentage of participants | 84.3 [62.5 to 93.9]

6. Other Pre Specified Outcome: Viability of Treatment
Description: Treatment is considered viable when the Study Device is removed and the structure is either resolved or improved without the need for re-stenting at the time of Study Device removal.
Time Frame: Upon Removal
Population: Subjects with stent removal data available
Measure: Count of Participants; unit: Participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 32
Participants | 26

7. Other Pre Specified Outcome: Secondary Patency Post Study Device Removal
Description: Secondary patency post study device removal is defined as the absence of stricture recurrence from time of Study Device removal to study completion or lost to follow up. Secondary Patency is also known as Long Term Stricture Resolution.
Time Frame: 15 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 33
percentage of participants | 67.8 [48.0 to 81.3]

8. Other Pre Specified Outcome: Primary Patency of Treated Stricture
Description: Primary patency of the treated stricture is defined as freedom from stricture intervention due to occlusion following Study Device removal.
Time Frame: 15 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE VIABIL
Number analyzed (Participants) | 33
percentage of participants | 64.8 [45.2 to 78.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for patients upto 12 Months of treatment period with the stent and upto 15 Months of post stent removal
Arm/Group | GORE VIABIL
All-Cause Mortality (participants affected / at risk) | 2/36
Serious Adverse Events (participants affected / at risk) | 19/36
Other Adverse Events (participants affected / at risk) | 6/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE VIABIL (N=36)
Recurrence of obstructive jaundice (Hepatobiliary disorders) | 5 (5)
Pancreatitis (Hepatobiliary disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Papillary hemorrhage (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 4 (4)
Other (General disorders) | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE VIABIL (N=36)
Other (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. Sponsor can require changes to the communication as necessary to ensure the proper use of any references to itself, its trademarks, and trade names and to correct inaccuracies in any technical specifications or descriptions of the device, including its component materials.